CLINICAL TRIAL: NCT06545682
Title: Phase Ib Study of AlpeliSib With PEmbroLizumab in Patients With mEtastatic Breast caNcer or melanomA (SELENA)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0173; NCI-2024-06339 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Melanoma (Skin Cancer); Breast Cancer; Brain Metastasases
MeSH Terms: conditions — Melanoma; Breast Neoplasms | interventions — Alpelisib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Study treatment will be administered on an outpatient basis.
  Interventions: Drug: Alpelisib + Pembrolizumab
- Dose Expansion (Experimental): Study treatment will be administered on an outpatient basis.
  Interventions: Drug: Alpelisib + Pembrolizumab

INTERVENTIONS:
Drug: Alpelisib + Pembrolizumab — Given by mouth (PO) Given by vein (IV)
  Other Names: BYL 719

SUMMARY:
To find a recommended dose of the combination of alpelisib and pembrolizumab that can be given to patients with metastatic breast cancer or melanoma.

DETAILED DESCRIPTION:
Primary Objective:

To determine the safety, tolerability, maximum tolerated dose (MTD), and/or recommended Phase II dose (RP2D) of the combination of alpelisib and pembrolizumab in patients with advanced/metastatic melanoma with and without brain metastasis and advanced/metastatic TNBC with brain metastasis.

Secondary Objectives:

To determine ORR as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 in all patients.

Exploratory Objectives:

To assess effects on exploratory biomarkers, including serum biomarkers, alterations in hematopoietic subpopulations as measured by multicolor flow cytometry and multimodal single cell analysis, and effects on the leukemic cells as assessed by gene panel analysis and/or single cell DNA-analysis.

To evaluate exposure by measuring PK.

To evaluate immunogenicity by assessing antidrug antibodies (ADA).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years or older.
2. Patients must be willing and able to provide informed consent.
3. In the dose escalation, patients must have histologically documented locally advanced, unresectable, or metastatic melanoma or TNBC that has progressed on treatments that are known to prolong survival or for which no standard treatment is available or refused such therapy. Presence of active brain metastases is not required. Patients with active metastases as defined below can be eligible in the dose escalation.
4. In the dose expansion, patients must have histologically documented locally advanced, unresectable, or metastatic melanoma or TNBC that has progressed on treatments that are known to prolong survival or for which no standard treatment is available or refused such therapy.

   1. Melanoma patients without brain metastases who have progressed on an anti-PD-1 or anti-PD-L1-based regimen.
   2. Melanoma patients with active and untreated brain metastases who have progressed on an anti-PD-1 or anti-PD-L1-based regimen.
   3. TNBC patients (defined as ER <1%, HER2 0, 1+, 2+, and fluorescence in situ hybridization negative) with active untreated brain metastases. Prior treatment with anti-PD-1/anti-PD-L1 is not required.
5. All patients must have had a brain magnetic resonance imaging (MRI) scan in the previous 28 days to confirm eligibility for the following cohorts:

   1. Dose escalation and dose expansion Cohort 1: Confirmed absence of untreated brain metastases in patients with histologically confirmed advanced melanoma. Prior surgery for brain metastases must have been completed at least 4 weeks prior study treatment initiation, whole brain radiation therapy must have been completed at least 3 weeks prior to study treatment initiation, and stereotactic radiosurgery must have been completed within 7 days prior to study treatment initiation.
   2. Dose escalation and dose expansion Cohorts 2 and 3: At least one confirmed measurable untreated brain lesion ≥ 0.5 cm and < 3.0 cm in the longest axis.
6. Has measurable disease based on the RECIST v1.1.
7. Has adequate organ function as defined in Table 2:
8. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Appendix 4).
9. Has a life expectancy of at least 12 weeks.
10. Able to swallow and retain orally administered medication.
11. In the dose expansion, patients with EC disease must be willing to provide tissue from a newly obtained, safely accessible core or excisional biopsy lesion at pre-treatment and at least one time point while on study treatment. Correlative biopsies will be optional in the dose escalation portion of the study. Newly obtained biopsy is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of study treatment on Day 1 without intervening systemic therapy.
12. Women of childbearing potential (WOCBP) should have a negative urine pregnancy test within 72 hours prior to receiving the first dose of study treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. Alpelisib and pembrolizumab can cause fetal harm when administered to a pregnant woman. Therefore, WOCBP must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from the time of screening through 4 months after the last dose of study treatment. Refer to Pregnancy Assessment Policy MD Anderson Cancer Center (MDACC) Institutional Policy # CLN1114. This includes all female patients between the onset of menses and 55 years unless the patient presents with an applicable exclusionary factor such as one of the following:

    1. Postmenopausal (no menses in ≥ 12 consecutive months)
    2. History of hysterectomy or bilateral salpingo-oophorectomy
    3. Ovarian failure (follicle-stimulating hormone and estradiol in menopausal range and have received whole pelvic radiation therapy)
    4. History of bilateral tubal ligation or another surgical sterilization procedure
14. Approved methods of birth control are as follows: hormonal contraception (i.e., birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device, tubal ligation or hysterectomy, patient/partner post vasectomy, implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the study and the study treatment washout period is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
15. Male patients with partner(s) of childbearing potential must agree to use adequate contraception from the time of screening through 4 months after the last dose of study treatment.

Exclusion Criteria:

1. Has a history of or active autoimmune disease, as follows: history of inflammatory bowel disease, history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]), motor neuropathy considered of autoimmune origin (e.g., Guillain-Barré syndrome and myasthenia gravis), or history of autoimmune thyroiditis (patients may be eligible if their current thyroid disorder is treated and stable with replacement or other medical therapy).
2. Has active infection or had a serious general medical condition(s) (such as vascular accident) in the past 6 months.
3. Any unresolved > Grade 1 toxicity (per CTCAE v5.0) from previous anticancer therapy or previously administered agent at the time of enrollment, except for alopecia and Grade 2 anemia (if hemoglobin is > 9 g/dL). Note: If the patient received major surgery, he/she must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
4. Patients who received chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to starting study treatment.
5. Presence of any clinically significant gastrointestinal abnormality or other condition(s) (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection) that may alter absorption such as malabsorption syndrome or major resection of the stomach or substantial portion of the small intestine based on investigator discretion.
6. Previous major surgery within 14 days prior to enrollment.
7. Evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, hepatic, renal, or cardiac disease).
8. Established diagnosis of diabetes mellitus type I or uncontrolled type II (based on fasting blood glucose and HbA1c [see inclusion criteria #4]).
9. History of acute pancreatitis within 1 year of screening or past medical history of chronic pancreatitis.
10. History of severe cutaneous reaction, such as SJS, erythema multiforme (EM), TEN, or drug reaction with eosinophilia and systemic symptoms (DRESS).
11. Based on average of triplicate 12-lead electrocardiogram (ECG), a mean resting QTc interval using Fridericia formula > 450 msec for males and > 470 msec for females at screening or a history of congenital long QT syndrome or QTc > 480 msec for patients with a bundle branch block.
12. History or evidence of cardiovascular risk including any of the following:

    1. History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, stenting, or bypass grafting within 6 months prior to enrollment.
    2. Class III or IV heart failure as defined by the New York Heart Association functional classification system.
    3. Known left ventricular ejection fraction < 50%.
    4. Known cardiac metastases.
13. Poorly controlled hypertension (defined as systolic blood pressure ≥150 mmHg or diastolic blood pressure >100 mmHg based on a mean of three measurements taken at approximately 2-minute intervals).

    Note: Initiation or adjustment of antihypertensive medication(s) is permitted if done 30 or more days prior to enrollment.
14. For dose expansion Cohorts 2 and 3 with active brain metastases:

    1. Patients must not have any of the following on the screening brain MRI:

       * Any untreated brain lesions > 3.0 cm in size.
       * Any brain lesion thought to require immediate local therapy, including (but not limited to) a lesion in an anatomic site where increase in size or possible treatment-related edema may pose risk to the patient (e.g., brainstem lesions). Patients who undergo local treatment for such lesions may still be eligible for the study.
    2. Ongoing use of systemic corticosteroids for control of symptoms of brain metastases at a total daily dose of dexamethasone (or equivalent) > 4 mg.

       * Poorly controlled (> 1/week) generalized or complex partial seizures, or manifestation of neurologic progression due to brain metastases notwithstanding CNS-directed therapy.
15. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorder that in the opinion of the treating physician or principal investigator (PI) would interfere with cooperation with the requirements of the trial.
18. Known history of hepatitis B or C or positive test for human immunodeficiency virus.
19. Has received a live vaccine within 30 days of planned start of study treatment.

    Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; COVID-19 vaccines are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
20. Current use of or anticipated requirement during the study of any prohibited medication(s) (See Section 5.5.2).
21. History of allergic reactions attributed to compounds of similar chemical or biologic composition to alpelisib and pembrolizumab.
22. Pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-08-03 (Estimated); Study Completion 2029-08-03 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ecaterina Dumbrava, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org